CLINICAL TRIAL: NCT05895084
Title: Neural Markers of Static & Dynamic Balance Before & After Yoga in Adults With Brain Injury
Brief Title: Neural Markers of Balance in Adults With Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECI Feasibility Study
Record Dates: First submitted 2023-03-31; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Yoga (Experimental): Yoga includes breath work (pranayama), gentle stretching and holding of postures (asanas), and meditation (dhyana). Modifications/adaptations are incorporated so all participants can successfully complete the yoga intervention. Yoga is delivered in a standardized progression, including: focused, slow breath with movement and breathwork throughout every session; mantras, progressively challenging yoga postures (sitting, standing, and floor); and meditation
  Interventions: Behavioral: Group Yoga

INTERVENTIONS:
Behavioral: Group Yoga — Yoga is delivered as described in an earlier section in a group format. Classes are an hour in duration and occur once per week for 8 weeks, and they are led by an adaptive yoga specialist.
  Other Names: Adaptive Yoga

SUMMARY:
The feasibility study is designed to assess the feasibility of conducting a group yoga intervention and acquiring neuroimaging data in adults with chronic brain injury.

DETAILED DESCRIPTION:
In the United States in 2014, nearly 2.9 million individuals sustained traumatic brain injuries that resulted in emergency department visits, hospitalizations, and death. Traumatic brain injury (TBI) is caused by trauma, or an external force that creates rapid acceleration and deceleration of the brain within the skull creating lasting neurophysiological dysfunction. Although there are many effective treatment strategies for the weeks and months post-injury (e.g. intensive, multi-disciplinary in-patient rehabilitation), millions of individuals are living with residual disability from brain injury following discharge to home. This residual disability can include significant social, cognitive, emotional, and physical impairment. To date, there are limited strategies for treating the residual deficits of chronic brain injury. One such physical deficit is balance impairment, which is associated with increased fall risk, reduced community integration, and decreased quality of life. The use of intensive, holistic rehabilitation may be effective for improving balance and other impairments in individuals with chronic brain injury. Yoga, a holistic treatment option, is thought to be more therapeutic than traditional exercise because of the integration of the mind, body, and spirit. Further, yoga can be modified to accommodate individual abilities and needs. And, unlike formal rehabilitation, yoga does not need to be approved by insurance or prescribed by a physician and adapted yoga is available in the community. Thus, yoga is readily available, so long as yoga instructors are trained to appropriately modify activities. Recently, the research team found that group yoga improved balance performance in seven adults with chronic brain injury. This study is designed to test the feasibility of conducting another group yoga intervention and acquiring neuroimaging data before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults, ages 18+
* Diagnosis of traumatic brain injury (TBI) or acquired brain injury (ABI) that occurred ≥ 6 months prior,
* Self-reported balance limitations.

Exclusion Criteria:

* Ability to engage in non-adapted (i.e. mainstream) yoga classes
* Standard contraindications for MRI (e.g. metal plates in head, claustrophobia, etc.)*

  * Individuals could still participate in the group yoga intervention even if they could not complete MRI scans.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Change in Balance Performance from Baseline to Post-Intervention Timepoint | Baseline was ~ 2 weeks before the start of group yoga; Post-Intervention was after the last group yoga class, which was 12-13 weeks after baseline assessment.
  Six balance tasks, adapted from the Berg Balance Scale, were administered with simultaneous functional near infrared spectroscopy (see secondary outcomes). Each balance task was evaluated using Functional Independence Measure (FIM) scoring, ranging from 0 (dependent, unable to do) to 7 (independent, able to do without help). A composite score was generated by averaging FIM scores from each balance task. Change in balance was quantified as the difference in the post-intervention balance composite score and the baseline balance composite score.
Change in Executive Functioning from Baseline to Post-Intervention Timepoint | Baseline was ~ 2 weeks before the start of group yoga; Post-Intervention was after the last group yoga class, which was 12-13 weeks after baseline assessment.
  Executive function was assessed with a self-report measure, the Behavior Rating Inventory of Executive Function - Adult Version. The BRIEF-A includes nine clinical scales: inhibit, self-monitor, plan/organize, shift, initiate, task monitor, emotional control, working memory and organization of materials. Items are self-rated using a three-point frequency scale (1 = never; 2=sometimes; 3=often). These items contribute to two broad indexes, behavioral regulation and metacognition, which are combined for a summary score. Raw scores are transformed into a T-score. Higher T scores reflect more reported problems and T scores at or above 65 are considered clinically significant.

SECONDARY OUTCOMES:
Resting State Functional Magnetic Resonance Imaging (rs-fMRI) - Feasibility Benchmark of Safety at Baseline | Baseline was ~ 2 weeks before the start of group yoga.
  The feasibility of safely acquiring rs-fMRI data was defined as the following: Detect 100% MRI contraindications during screening. Sustain zero instances of adverse events (e.g. pain or significant anxiety) or falls during data acquisition.
Resting State Functional Magnetic Resonance Imaging (rs-fMRI) - Feasibility Benchmark of Safety at Post-Intervention | Post-Intervention was after the last group yoga class, which was 12-13 weeks after baseline assessment.
  The feasibility of safely acquiring rs-fMRI data was defined as the following: Detect 100% MRI contraindications during screening. Sustain zero instances of adverse events (e.g. pain or significant anxiety) or falls during data acquisition.
Resting State Functional Magnetic Resonance Imaging (rs-fMRI) - Feasibility Benchmark of Data Quality at Baseline | Baseline was ~ 2 weeks before the start of group yoga.
  Rs-fMRI data quality was defined as meeting the following: Achieve time series quality indices < 3.5 * median absolute deviation (MAD) in ≥ 80% of data time points. Observe similar quality indices as achieved in a normative sample.
Resting State Functional Magnetic Resonance Imaging (rs-fMRI) - Feasibility Benchmark of Data Quality at Post Intervention | Post-Intervention was after the last group yoga class, which was 12-13 weeks after baseline assessment.
  Rs-fMRI data quality was defined as meeting the following: Achieve time series quality indices < 3.5 * median absolute deviation (MAD) in ≥ 80% of data time points. Observe similar quality indices as achieved in a normative sample.
Functional Near-Infrared Spectroscopy (fNIRS) - Feasibility Benchmark of Safety at Baseline | Baseline was ~ 2 weeks before the start of group yoga.
  The feasibility of safely acquiring fNIRS data was defined as the following: Have zero instances of adverse events (e.g. pain or anxiety) or falls during data acquisition.
Functional Near-Infrared Spectroscopy (fNIRS) - Feasibility Benchmark of Safety at Post-Intervention. | Post-Intervention was after the last group yoga class, which was 12-13 weeks after baseline assessment.
  The feasibility of safely acquiring fNIRS data was defined as the following: Have zero instances of adverse events (e.g. pain or anxiety) or falls during data acquisition.
Functional Near-Infrared Spectroscopy (fNIRS) - Feasibility Benchmark of Data Quality at Baseline | Baseline was ~ 2 weeks before the start of group yoga.
  FNIRS data quality was defined as meeting the following: Reach acceptable signal optimization and quality levels in ≥ 80% of participants assessed. Successfully detect and remove motion artifacts from data in ≥ 80% of participants assessed.
Functional Near-Infrared Spectroscopy (fNIRS) - Feasibility Benchmark of Data Quality at Post-Intervention | Post-Intervention was after the last group yoga class, which was 12-13 weeks after baseline assessment.
  FNIRS data quality was defined as meeting the following: Reach acceptable signal optimization and quality levels in ≥ 80% of participants assessed. Successfully detect and remove motion artifacts from data in ≥ 80% of participants assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn A Stephens, PhD, OTR/L, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University - SCORE Research Lab, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data can be acquired upon request to the study PI, Dr. Jaclyn Stephens.
Supporting Information: Study Protocol, SAP
Time Frame: Upon request - available for 5 years